CLINICAL TRIAL: NCT02164240
Title: A Non-randomized, Open-label Phase Ib Study of SUnitinib Alternating With REgorafenib in Patients With Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (GIST) Progressing After Prior Therapy With Tyrosine Kinase Inhibitors
Brief Title: Phase Ib Study of SUnitinib Alternating With REgorafenib in Patients With Metastatic and/or Unresectable GIST
Acronym: SURE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bayer (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Suzanne George, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-149
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib alternated with Regorafenib (Experimental): The treatment cycle is defined as 28 days. Treatment consists of 3 days of once daily sunitinib alternating with 4 days of once daily regorafenib throughout each cycle. The starting dose level is sunitinib 37.5 mg/d and regorafenib 120 mg/d, and doses will be escalated in subsequent cohorts following a classical 3+3 design up to sunitinib 50 mg/d and regorafenib 160 mg/d or until maximum tolerable dosage and recommended phase II dose is determined. An alternative scheme of 4-week cycles of the same regimen but with 21 days of dosing followed by 7 days of rest will be studied in case of toxicities during d 22-28 of the starting 4-weeks continuous cycles. Tumor assessments performed at baseline and after every two dosing cycles to assess response. Toxicity monitored throughout the study.
  Interventions: Drug: Sunitinib; Drug: Regorafenib

INTERVENTIONS:
Drug: Sunitinib — Intervention Description: 3 days of once daily sunitinib alternating with 4 days of once daily regorafenib throughout each 28 day cycle. The starting dose level (level 1) is sunitinib 37.5 mg/d and regorafenib 120 mg/d, and doses will be escalated in subsequent cohorts following a classical 3+3 design up to sunitinib 50 mg/d and regorafenib 160 mg/d or until maximum tolerable dosage (MTD) and recommended phase II dose (RP2D) is determined. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Sutent
Drug: Regorafenib — Intervention Description: 3 days of once daily sunitinib alternating with 4 days of once daily regorafenib throughout each 28 day cycle. The starting dose level (level 1) is sunitinib 37.5 mg/d and regorafenib 120 mg/d, and doses will be escalated in subsequent cohorts following a classical 3+3 design up to sunitinib 50 mg/d and regorafenib 160 mg/d or until maximum tolerable dosage (MTD) and recommended phase II dose (RP2D) is determined. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Stivarga

SUMMARY:
The purpose of this research study is to determine the safety and tolerability of sunitinib alternating with regorafenib in participants with advanced gastrointestinal stromal tumor GIST, if the standard approved therapies (imatinib, sunitinib and regorafenib) have failed to control the disease. Additionally, this study seeks to determine the highest dose that can be given safely for this combination of drugs.

DETAILED DESCRIPTION:
This is a non-randomized, open label, single-center, single-arm, phase Ib study to evaluate the safety and the preliminary efficacy of short cycles of sunitinib alternated with regorafenib in participants with metastatic and/or unresectable gastrointestinal stromal tumor GISTs with prior failure of tyrosine kinase inhibitors (TKI). The study consists of two cohorts: a dose-escalation, dose-finding cohort, and dose-expansion cohort. Between 6 to 15 patients are expected to be included in the escalation cohort. A total of 20 eligible and evaluable patients will be included in the expansion cohort to further assess toxicity and evaluate preliminary efficacy.

Each treatment cycle lasts 28 days (4 weeks), during which time you will be taking the study drug, sunitinib, for the first 3 days of the week, followed by the study drug, regorafenib, for the last 4 days of the week. The study drugs will be taken continuously for 4 weeks each cycle, unless the study team instructs you otherwise. Each participant will receive a study diary. The diary will also include special instructions for taking the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of study entry.
* Histologically confirmed metastatic and/or unresectable GIST. Patients must demonstrate prior failure to at least imatinib, sunitinib and regorafenib (4th line and beyond). Any number of previous therapies for GIST is allowed.
* Measurable disease per modified RECIST 1.1. A lesion in a previously irradiated area is ineligible to be considered as measurable disease unless there is objective evidence of progression of the lesion prior to study enrollment.
* ECOG performance status 0 or 1 (see Appendix A).
* Participants must have adequate organ and marrow function as outlined in the protocol.
* Patients must be able to swallow oral medication.
* Willingness to use effective means of birth control throughout the duration of clinical study and for at least 3 months after completion of study drug.
* Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of study drug administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Use of any approved tyrosine kinase inhibitors or investigational agents within 2 weeks or 6 half-lives of the agent, whichever is shorter, prior to receiving study drugs.
* Patients with intolerance to sunitinib and/or regorafenib.
* Participants who have had radiotherapy within 4 weeks prior to study entry.
* Major surgery, or significant traumatic injury within 4 weeks prior to study entry.
* Presence of symptomatic or uncontrolled brain or central nervous system metastases.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Individuals with a history of a different malignancy, other than cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy OR other primary malignancy is neither currently clinically significant nor requiring active intervention.
* Clinically significant cardiac arrhythmias and/or patients who require anti-arrhythmic therapy (excluding beta blockers or digoxin). Patients with controlled atrial fibrillation are not excluded.
* History of clinically significant cardiac disease or congestive heart failure > NYHA class 2 (See Appendix C). Patients must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months.
* Hypertension as defined by systolic blood pressure >140 mmHg or diastolic blood pressure > 90 mmH despite optimal medical management.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than 1 month before the start of study medication).
* Patients with evidence or history of any bleeding diathesis, irrespective of severity.
* Ongoing infection ≥ Grade 2.
* Patients with any seizure disorder requiring medication.
* Non-healing wound, ulcer, or bone fracture.
* Persistent proteinuria Grade 2 or higher measured by urine protein:creatinine ratio on a urine sample or during 24-hour assessment.
* HIV-positive individuals on combination antiretroviral therapy.
* Patients with active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Uncontrolled intercurrent illness.
* Pregnant or lactating females.
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol.
* Strong CYP3A4 inhibitors within 28 days or 5 drug half-lives, whichever is longer, before start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Serrano C, Leal A, Kuang Y, Morgan JA, Barysauskas CM, Phallen J, Triplett O, Marino-Enriquez A, Wagner AJ, Demetri GD, Velculescu VE, Paweletz CP, Fletcher JA, George S. Phase I Study of Rapid Alternation of Sunitinib and Regorafenib for the Treatment of Tyrosine Kinase Inhibitor Refractory Gastrointestinal Stromal Tumors. Clin Cancer Res. 2019 Dec 15;25(24):7287-7293. doi: 10.1158/1078-0432.CCR-19-2150. Epub 2019 Aug 30. PMID 31471313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The "Protocol Enrollment" number reflects the 14 participants who completed the informed consent process, were determined eligible following screening, and were registered in the protocol registration system per study protocol. The "Started in Participant Flow" number reflects the 13 participants who started on the course of study drug treatment following registration (1 of the 14 enrolled participants did not).
Groups:
- Sunitinib 37.5 and Regorafenib 120; Expansion Sunitinib 37.5 Regorafenib 120: Patients were enrolled and treated with sunitinib 37.5mg daily alternating with regorafenib 120mg daily
- Sunitinib 37.5 and Regorafenib 160: Patients were enrolled and treated with sunitinib 37.5mg daily alternating with regorafenib 160mg daily
Period: Overall Study
Arm/Group | Sunitinib 37.5 and Regorafenib 120 | Sunitinib 37.5 and Regorafenib 160 | Expansion Sunitinib 37.5 Regorafenib 120
Started | 4 | 5 | 4
Completed | 4 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who received treatment were included in the analysis
Groups:
- Sunitinib Alternated With Regorafenib: Sunitinib: Intervention Description: 3 days of once daily sunitinib alternating with 4 days of once daily regorafenib throughout each 28 day cycle.
Arm/Group | Sunitinib Alternated With Regorafenib
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 63.5 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Dose-escalation cohort is to determine the frequency and characteristics of DLTs of alternation of sunitinib and regorafenib at each dose level during the first cycle of therapy. Toxicity will be graded accordingly with NCI CTCAE version 4.0
Time Frame: Up to Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Sunitinib 37.5 and Regorafenib 120: Patients were enrolled and treated with sunitinib 37.5 mg daily alternating with regorafenib 120mg daily
- Sunitinib 37.5 and Regorafenib 160: patients were enrolled and treated with sunitinib 37.5 mg daily and regorafenib 160mg daily
- Expansion Sunitinib 37.5 Regorafenib 120: RPD2 determined to be sunitinib 37.5mg daily and regorafenib 120mg daily and therefore, per protocol, the cohort was expanded at this dose level
Arm/Group | Sunitinib 37.5 and Regorafenib 120 | Sunitinib 37.5 and Regorafenib 160 | Expansion Sunitinib 37.5 Regorafenib 120
Number analyzed (Participants) | 4 | 5 | 4
Participants | 4 | 5 | 4

2. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Percentage of participants who experienced complete response, partial response or stable disease per RECIST 1.1 at 16 weeks
Time Frame: 16 weeks
Population: clinical benefit was analyzed across the entire population based on the pre-planned study design
Measure: Count of Participants; unit: Participants
Groups:
- Sunitinib and Regorafenib: Patients were enrolled and treated with sunitinib alternating with regorafenib
Arm/Group | Sunitinib and Regorafenib
Number analyzed (Participants) | 13
Participants | 0
Statistical Analysis 1: Comparison: Sunitinib and Regorafenib; Clinical benefit rate of at least 30% at 16 weeks for the entire, combined population, was considered worthy of further study; Test type: Other; descriptive statistics only; Clinical Benefit Rate = 0, 95% CI 2-sided [0 to 24.7]

3. Secondary Outcome: Median Progression Free Survival (mPFS)
Description: Non-parametric Kaplan-Meier analysis to assess median progression free survival (mPFS)
Time Frame: From date of registration until date of protocol-defined progression while on this protocol, assessed up to 6 months
Population: all patients enrolled were analyzed as a single cohort for this endpoint based on pre-planned study design
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib and Regorafenib
Number analyzed (Participants) | 13
months | 1.9 [1.4 to 3.6]

ADVERSE EVENTS:
Groups:
- Cohort 1: SuRe120; Cohort 3: ExpSuRe120: Patients were enrolled and treated with sunitinib 37.5mg/d alternating with regorafenib 120 mg/d
- Cohort 2: SuRe160: Patients were enrolled and treated with sunitinib 37.5mg/d alternating with regorafenib 160 mg/d
Arm/Group | Cohort 1: SuRe120 | Cohort 2: SuRe160 | Cohort 3: ExpSuRe120
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/5 | 2/4
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SuRe120 (N=4) | Cohort 2: SuRe160 (N=5) | Cohort 3: ExpSuRe120 (N=4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SuRe120 (N=4) | Cohort 2: SuRe160 (N=5) | Cohort 3: ExpSuRe120 (N=4)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 4 | 4 | 4
Pain (General disorders) | 0 | 0 | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 1
Weight loss (Investigations) | 2 | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Flushing (Vascular disorders) | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No